CLINICAL TRIAL: NCT01890018
Title: Partners and Alerts: A Study of Social Forces in Medication Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: 817167; 1C1CMS331009-01-00 (Other Grant/Funding Number: Center for Medicare & Medicaid Innovation (CMMI))
Record Dates: First submitted 2013-05-09; First posted 2013-07-01 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Acute Myocardial Infarction (AMI)
Keywords: Acute Myocardial Infarction (AMI); taking a statin medication; also have a medication adherence ratio (MPR)

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control (Active Comparator): This arm will use GlowCaps to have their adherence tracked with no additional modifications:
  Arm 1. Control group no modifications
  Electronic Pill Bottle tracking
  Interventions: Behavioral: Electronic Pill Bottle tracking
- Feedback group (Experimental): This arm will use GlowCaps to have their adherence tracked with the following modifications:
  Arm 2. Feedback group participants will receive an adherence message after 48 hours of not using the GlowCaps
  Electronic Pill Bottle tracking; Adherence Messaging
  Interventions: Behavioral: Electronic Pill Bottle tracking; Behavioral: Adherence Messaging
- Adherence partner group (Experimental): This arm will use GlowCaps to have their adherence tracked with the following modifications:
  Arm 3. Adherence partner group participants will designate a family member or friend who will serve as an adherence partner, encouraging adherence of the patient
  Electronic Pill Bottle tracking; Social Influence
  Interventions: Behavioral: Electronic Pill Bottle tracking; Behavioral: Social Influence
- Adherence partner along with feedback (Experimental): This arm will use GlowCaps to have their adherence tracked with the following modifications:
  Arm 4. Adherence partner along with feedback group participants will designate a family member or friend who will serve as an adherence partner, encouraging adherence of the patient, both the patient and partner will receive a message after 48 hours of not using the GlowCaps
  Electronic Pill Bottle tracking; Adherence Messaging; Social Influence
  Interventions: Behavioral: Electronic Pill Bottle tracking; Behavioral: Adherence Messaging; Behavioral: Social Influence

INTERVENTIONS:
Behavioral: Electronic Pill Bottle tracking — All 4 groups will use the GlowCaps, a remote monitoring bottle, to take their statin medications
Behavioral: Adherence Messaging — Some arms will receive adherence messages if they have not used the Glowcap bottles for 2 of the last 3 days.
  Arms: Adherence partner along with feedback; Feedback group
Behavioral: Social Influence — Some arms will select their own adherence feedback partner who will provide support in taking their medication as scheduled.
  Arms: Adherence partner along with feedback; Adherence partner group

SUMMARY:
The overall objectives of this study are to improve medication adherence of patients and subsequent health outcomes.

This study is designed to examine the existence of strong associations between social networks and health behavior. This study intends to demonstrate that social forces are particularly effective at building enduring habits for healthy behavior, specifically adherence to statin medication for this study. The investigators believe the improved medication adherence will result in fewer additional vascular events, following the most recent of these events, and will result in fewer patient hospitalizations. The investigators will leverage insights from the fields of social comparison (being provided with information about the actions of others prompts social comparison that can significantly influence behavior), social pressures (encouragement or discouragement from others is a powerful social force that can influence individual behavior), and social triggers (cues in the environment can motivate people to take certain actions and have powerful effects on purchasing behavior).

The results of this study and experience gained from the implementation of these interventions will be used to inform new versions of a larger trial intervention to be tested in new patient cohorts in a rapid cycle framework.

DETAILED DESCRIPTION:
This study is a 4-arm pilot study involving 248 patients (62 per arm) who are on a once-a-day statin who have a medication adherence ratio (MPR) that is less than 80%. Patients in all arms would receive a GlowCap, manufactured by Vitality Inc., which records pill-bottle openings and be asked to use the GlowCap for that medication for the duration of the study.

The study arms leverage two strategies that the investigators think will be particularly effective at improving adherence and may be even more effective when used in tandem. Patients in some arms will be asked to select an adherence partner: another person who can help them adhere to their medication regimen. The investigators will contact this adherence partner and ask them to officially accept this role and provide guidance of their choosing as to how they can help the patient adhere. In addition, patients in some arms will receive an alert whenever two full days pass without their GlowCap being opened (i.e. 48 hours of non-adherence). This alert will encourage them to begin taking their medication again. The design allows for some patients to have both an adherence partner and to receive alerts after 48 hours of non-adherence. In these arms, the adherence partner would also receive the alert after 48 hours of non-adherence. This introduces a two-by-two design.

Subjects would spend 6 months in their randomly assigned treatment, and the investigators will compare adherence of subjects in each of the arms to one another.

The investigators plan to track daily adherence of patients to a prescribed chronic disease drug using a new technology that electronically monitors when a pill bottle has been opened. In our control condition, patients will be monitored but not be provided with any reminders, adherence information, or inclusion of friend of family member to help them adhere to their medication. Our four additional treatments will either: (1) email the patient after 48 hours of non-adherence; (2) allow the patient to select friend or family member to encourage medication adherence; (3) email the patient, as well as patient-selected friends or family members after 48 hours of non-adherence; or (4) provide the patient with a daily email, text message, or phone call reminder to take the pill.

ELIGIBILITY:
Inclusion Criteria:

Patients must have

* experienced an AMI and have been placed on a once-a-day statin and have a medication adherence ratio (MPR) that is less than 80%.
* access to internet to create an account on Way to Heath.

Exclusion Criteria:

* There are no exclusion criterial for patients able to provide consent and who meet the eligibility criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Glowcap bottle openings/Medication Adherence | 6 months
  Primary outcome will measure the the number of days the GlowCap pill bottle is opened at least 1 time over the 6 month enrollment period, to be measured at 6 months after enrollment for each participant. Medication adherence for this study is considered to be at least 1 registered GlowCap opening for each day enrolled on the study. (N days at least 1 opening/180 days = Medication Adherence %)

SECONDARY OUTCOMES:
Patient pharmacy benefits-this will be a composite outcome measure assessing MPR | 18 months
  Secondary outcomes will be gap ratios and medication possession ratios.
Patient Claims records - this will be a composite outcome measure assessing frequency of hospitalization | 18 months
  Secondary outcomes will be the number of repeat vascular events, following a similar approach to MI-FREEE, hospitalization, repeat or new cardiovascular procedures, and cost.

CONTACTS AND LOCATIONS:
Overall Officials: Judd B Kessler, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Palmer MJ, Machiyama K, Woodd S, Gubijev A, Barnard S, Russell S, Perel P, Free C. Mobile phone-based interventions for improving adherence to medication prescribed for the primary prevention of cardiovascular disease in adults. Cochrane Database Syst Rev. 2021 Mar 26;3(3):CD012675. doi: 10.1002/14651858.CD012675.pub3. PMID 33769555
- [Derived] Kessler JB, Troxel AB, Asch DA, Mehta SJ, Marcus N, Lim R, Zhu J, Shrank W, Brennan T, Volpp KG. Partners and Alerts in Medication Adherence: A Randomized Clinical Trial. J Gen Intern Med. 2018 Sep;33(9):1536-1542. doi: 10.1007/s11606-018-4389-7. Epub 2018 Mar 15. PMID 29546659